CLINICAL TRIAL: NCT07203144
Title: Selenium Supplementation for Improving Depression in Children and Adolescents: Efficacy and Mechanistic Study
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Xinyu Zhou, professor, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1stChongqingMU---ZXY
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Depression - Major Depressive Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluoxetine combined with selenium yeast therapy (Experimental): In this group, participants will receive standard fluoxetine treatment along with adjunctive selenium yeast supplementation at a daily dose of 60-200 μg, aiming to investigate the role and mechanisms of selenium yeast in fluoxetine therapy.
  Interventions: Drug: selenium yeast supplementation
- Fluoxetine combined with placebo therapy (Placebo Comparator): Participants in this group, in addition to receiving conventional fluoxetine treatment, were administered 60-200 µg per day of a placebo identical in appearance and odor to selenium yeast as adjunctive therapy. The aim was to investigate the role of selenium yeast in fluoxetine treatment and to clarify whether it enhances the therapeutic effect.
  Interventions: Drug: Placebo yeast supplementation

INTERVENTIONS:
Drug: selenium yeast supplementation — In this intervention, patients will receive adjunctive selenium yeast supplementation at a daily dose of 60-200 μg in addition to fluoxetine. Symptom rating scales, biospecimen collection, and brain MRI will be conducted at baseline, week 4, and week 8 to investigate the adjunctive role of selenium in fluoxetine treatment for depression.
  Arms: Fluoxetine combined with selenium yeast therapy
Drug: Placebo yeast supplementation — In this intervention, patients will receive standard fluoxetine treatment combined with placebo yeast supplementation (60-200 μg/day), which is identical in appearance and odor to selenium yeast. The aim is to clarify the specific role of selenium in the treatment of depression.
  Arms: Fluoxetine combined with placebo therapy

SUMMARY:
The purpose of this study is to investigate the role and mechanisms of selenium in depression among children and adolescents, aiming to provide new insights for understanding the pathogenesis and treatment of depression in this population.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled trial will evaluate the efficacy and safety of selenium supplementation (selenium yeast) combined with fluoxetine in children and adolescents with major depressive disorder (MDD). Eligible participants are aged [specific age range if applicable], meet DSM-5 criteria for a current depressive episode, and have a CDRS-R score ≥40 confirmed by trained psychiatrists. A total of [planned sample size] participants will be randomized 1:1 to receive either fluoxetine plus selenium yeast or fluoxetine plus placebo. Selenium yeast will be administered at 60-200 μg/day. Fluoxetine will begin at 10 mg/day and may be adjusted by the treating psychiatrist within a range of 20-60 mg/day. The placebo consists of commercially available yeast tablets identical in appearance, taste, and size to selenium yeast, administered at 60-200 μg/day. Biological samples (blood, urine, stool) will be collected for routine laboratory tests, thyroid, liver, and kidney function, and serum will be analyzed for selenium and ferroptosis-related biomarkers. Brain MRI will also be performed. These assessments will be repeated at weeks 4 and 8 of treatment, together with rating scale evaluations and biospecimen collection. The primary outcome is the change in depressive symptoms, measured by the CDRS-R and Beck Depression Inventory (BDI). Secondary outcomes include anxiety symptoms (SCARED, HAMA), overall clinical improvement (CGI-S, CGI-I), manic symptoms (YMRS), suicide risk (C-SSRS), quality of life (PedsQL 4.0), sleep quality (PSQI), and rumination (RSS). Safety will be monitored through adverse events, vital signs, laboratory tests, and tolerability assessments. This study will provide preliminary evidence on the adjunctive role of selenium supplementation in fluoxetine treatment for adolescent depression and inform future large-scale trials.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12-18 years;
* Diagnosed with major depressive disorder according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), using the K-SADS-PL diagnostic tool;
* A score of ≥28 on the Children's Depression Rating Scale-Revised (CDRS-R);
* Adequate visual and auditory abilities to complete the study;
* Willingness to participate in the study with informed consent signed by both the participant and a legal guardian.

Exclusion Criteria:

* Patients with severe psychiatric disorders such as bipolar disorder, schizophrenia, bulimia nervosa, anorexia nervosa, or primary obsessive-compulsive disorder;
* Those with severe physical illnesses or other life-threatening conditions; patients in a current depressive episode with a clear suicidal plan or history of suicide attempt;
* Individuals with a history of substance or drug abuse;
* Those requiring immediate hospitalization for psychiatric disorders;
* Patients currently taking medications contraindicated with the investigational drug or that may interfere with its efficacy;
* Those who have received modified electroconvulsive therapy (MECT) within the past 12 months;
* Individuals allergic to selenium yeast protein, including those with allergic rhinitis, gastrointestinal sensitivity, allergic constitution, or autoimmune diseases such as Graves' disease or Hashimoto's thyroiditis;
* Patients with contraindications to magnetic resonance imaging (MRI);
* Aand left-handed individuals.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 172 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in CDRS-R (Children's Depression Rating Scale) scores from baseline | Week 4 and Week 8 of treatment
  The Children's Depression Rating Scale-Revised (CDRS-R) has a minimum score of 17 and a maximum score of 113. Higher scores indicate greater severity of depression.
  Primary Outcome Measure is clinical response (≥ 50% reduction in CDRS-R scores from baseline)；

SECONDARY OUTCOMES:
Change in BDI-II (Baker Depression Scale) scores from baseline | Week 4 and Week 8 of treatment
  The BDI-II (Beck Depression Inventory-II) is a self-report scale for assessing depression, with a minimum score of 0 and a maximum score of 63. Higher scores indicate more severe depression. One of the secondary outcome measures is the change in the BDI-II score compared to the baseline.
Change in SCARED (The Screen for Child Anxiety-Related Emotional Disorders) scores from baseline | Week 4 and Week 8 of treatment
  The SCARED (Screen for Child Anxiety-Related Emotional Disorders) is a self-report scale used to assess anxiety symptoms. The minimum score is 0 and the maximum score is 82, with higher scores indicating more severe anxiety. One of the secondary outcome measures is the improvement in anxiety, represented by the change in the SCARED score compared to the baseline.
Change in suicide risk from baseline on the C-SSRS (Columbia Suicide Severity Rating Scale) | Week 4 and Week 8 of treatment
  The Columbia Suicide Severity Rating Scale (C-SSRS) is a tool used to assess the risk of self-harm or suicide, and it does not have a score. One of the secondary outcome measures is to evaluate whether there is an improvement in self-harm or suicidal ideation and behavior compared to the baseline.
Change in PSQI (Pittsburgh Sleep Quality Index) scores from baseline | Week 4 and Week 8 of treatment
  The PSQI (Pittsburgh Sleep Quality Index) is a self-report scale used to assess sleep quality. The minimum score is 0, and the maximum score is 60. Higher scores indicate poorer sleep quality. One of the secondary outcome measures is to evaluate the change in the PSQI score compared to the baseline, assessing whether sleep treatment has led to improvement.
Change in PedsQL4.0 (The Pediatric Quality of Life Inventory) scores from baseline | Week 4 and Week 8 of treatment
  The PedsQL 4.0 (The Pediatric Quality of Life Inventory) is a self-report scale used to assess the quality of life in children. The minimum score is 0, and the maximum score is 92. Higher scores indicate better quality of life. One of the secondary outcome measures is the change in the PedsQL score compared to the baseline, assessing whether there has been an improvement in quality of life.
Change in CGI-S (Clinical Global Impressions-Severity Scales) scores from baseline | Week 4 and Week 8 of treatment
  Improvement in overall clinical impression severity ( 7-point scale, with 1 being normal and 7 being among the most severely damaged )
Change in CGI-I (Clinical Global Impressions-Improvement Scales) scores from baseline | Week 4 and Week 8 of treatment
  Improvement of clinical general Impression scale (7-point scale,7 denoting a very significant deterioration)
Change in RSS (Ruminative Responses Scale) | Week 4 and Week 8 of treatment
  The level of improvement in negative thinking(The minimum score is 22 and the maximum score is 88; the higher the total score, the more reflective thinking the more severe it is).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Result] Barker MM, Beresford B, Bland M, Fraser LK. Prevalence and Incidence of Anxiety and Depression Among Children, Adolescents, and Young Adults With Life-Limiting Conditions: A Systematic Review and Meta-analysis. JAMA Pediatr. 2019 Sep 1;173(9):835-844. doi: 10.1001/jamapediatrics.2019.1712. PMID 31282938
- [Result] Hankin BL. Depression from childhood through adolescence: Risk mechanisms across multiple systems and levels of analysis. Curr Opin Psychol. 2015 Aug;4:13-20. doi: 10.1016/j.copsyc.2015.01.003. PMID 25692174
- [Result] Consoli A, Peyre H, Speranza M, Hassler C, Falissard B, Touchette E, Cohen D, Moro MR, Revah-Levy A. Suicidal behaviors in depressed adolescents: role of perceived relationships in the family. Child Adolesc Psychiatry Ment Health. 2013 Mar 16;7(1):8. doi: 10.1186/1753-2000-7-8. PMID 23497551
- [Result] Dolle K, Schulte-Korne G. The treatment of depressive disorders in children and adolescents. Dtsch Arztebl Int. 2013 Dec 13;110(50):854-60. doi: 10.3238/arztebl.2013.0854. PMID 24399027
- [Result] Cipriani A, Zhou X, Del Giovane C, Hetrick SE, Qin B, Whittington C, Coghill D, Zhang Y, Hazell P, Leucht S, Cuijpers P, Pu J, Cohen D, Ravindran AV, Liu Y, Michael KD, Yang L, Liu L, Xie P. Comparative efficacy and tolerability of antidepressants for major depressive disorder in children and adolescents: a network meta-analysis. Lancet. 2016 Aug 27;388(10047):881-90. doi: 10.1016/S0140-6736(16)30385-3. Epub 2016 Jun 8. PMID 27289172
- [Result] Kryukov GV, Castellano S, Novoselov SV, Lobanov AV, Zehtab O, Guigo R, Gladyshev VN. Characterization of mammalian selenoproteomes. Science. 2003 May 30;300(5624):1439-43. doi: 10.1126/science.1083516. PMID 12775843
- [Result] Rayman MP. Selenium and human health. Lancet. 2012 Mar 31;379(9822):1256-68. doi: 10.1016/S0140-6736(11)61452-9. Epub 2012 Feb 29. PMID 22381456
- [Result] Dang R, Wang M, Li X, Wang H, Liu L, Wu Q, Zhao J, Ji P, Zhong L, Licinio J, Xie P. Edaravone ameliorates depressive and anxiety-like behaviors via Sirt1/Nrf2/HO-1/Gpx4 pathway. J Neuroinflammation. 2022 Feb 7;19(1):41. doi: 10.1186/s12974-022-02400-6. PMID 35130906
- [Result] Xu C, Xiong Q, Tian X, Liu W, Sun B, Ru Q, Shu X. Alcohol Exposure Induces Depressive and Anxiety-like Behaviors via Activating Ferroptosis in Mice. Int J Mol Sci. 2022 Nov 10;23(22):13828. doi: 10.3390/ijms232213828. PMID 36430312
- [Result] Reeves MA, Hoffmann PR. The human selenoproteome: recent insights into functions and regulation. Cell Mol Life Sci. 2009 Aug;66(15):2457-78. doi: 10.1007/s00018-009-0032-4. Epub 2009 Apr 28. PMID 19399585
- [Result] Ferreira de Almeida TL, Petarli GB, Cattafesta M, Zandonade E, Bezerra OMPA, Tristao KG, Salaroli LB. Association of Selenium Intake and Development of Depression in Brazilian Farmers. Front Nutr. 2021 May 20;8:671377. doi: 10.3389/fnut.2021.671377. eCollection 2021. PMID 34095192
- [Result] Mokhber N, Namjoo M, Tara F, Boskabadi H, Rayman MP, Ghayour-Mobarhan M, Sahebkar A, Majdi MR, Tavallaie S, Azimi-Nezhad M, Shakeri MT, Nematy M, Oladi M, Mohammadi M, Ferns G. Effect of supplementation with selenium on postpartum depression: a randomized double-blind placebo-controlled trial. J Matern Fetal Neonatal Med. 2011 Jan;24(1):104-8. doi: 10.3109/14767058.2010.482598. Epub 2010 Jun 8. PMID 20528216
- [Result] Islam MR, Islam MR, Shalahuddin Qusar MMA, Islam MS, Kabir MH, Mustafizur Rahman GKM, Islam MS, Hasnat A. Alterations of serum macro-minerals and trace elements are associated with major depressive disorder: a case-control study. BMC Psychiatry. 2018 Apr 10;18(1):94. doi: 10.1186/s12888-018-1685-z. PMID 29631563
- [Result] Wang H, Jin M, Xie M, Yang Y, Xue F, Li W, Zhang M, Li Z, Li X, Jia N, Liu Y, Cui X, Hu G, Dong L, Wang G, Yu Q. Protective role of antioxidant supplementation for depression and anxiety: A meta-analysis of randomized clinical trials. J Affect Disord. 2023 Feb 15;323:264-279. doi: 10.1016/j.jad.2022.11.072. Epub 2022 Nov 25. PMID 36442656
- [Result] Albrakati A, Alsharif KF, Al Omairi NE, Alsanie WF, Almalki ASA, Abd Elmageed ZY, Elshopakey GE, Lokman MS, Bauomy AA, Abdel Moneim AE, Kassab RB. Neuroprotective Efficiency of Prodigiosins Conjugated with Selenium Nanoparticles in Rats Exposed to Chronic Unpredictable Mild Stress is Mediated Through Antioxidative, Anti-Inflammatory, Anti-Apoptotic, and Neuromodulatory Activities. Int J Nanomedicine. 2021 Dec 30;16:8447-8464. doi: 10.2147/IJN.S323436. eCollection 2021. PMID 35002238
- [Result] Beardslee WR, Brent DA, Weersing VR, Clarke GN, Porta G, Hollon SD, Gladstone TR, Gallop R, Lynch FL, Iyengar S, DeBar L, Garber J. Prevention of depression in at-risk adolescents: longer-term effects. JAMA Psychiatry. 2013 Nov;70(11):1161-70. doi: 10.1001/jamapsychiatry.2013.295. PMID 24005242